CLINICAL TRIAL: NCT00786942
Title: Bone Graft Necessity in Opening-Wedge High Tibial Osteotomy. A Randomized Clinical Trial
Brief Title: Bone Graft Necessity in Opening-Wedge High Tibial Osteotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Alessandro Rozim Zorzi, Unicamp
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Puddu
Record Dates: First submitted 2008-11-05; First posted 2008-11-06 (Estimated); Last update posted 2010-05-24 (Estimated); Status verified 2010-05

CONDITIONS: Osteoarthritis
Keywords: osteotomy; knee; varus deformity; bone graft
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): autologous bone graft
  Interventions: Procedure: high tibial osteotomy
- 2 (Experimental): without bone graft
  Interventions: Procedure: higi tibial osteotomy

INTERVENTIONS:
Procedure: high tibial osteotomy — addition of bone graft to fill the osteotomy gap
  Other Names: opening-wedge higi tibial osteotomy
  Arms: 1
Procedure: higi tibial osteotomy — the gap of the tibia is unfilled
  Other Names: opening-wedge higi tibial osteotomy
  Arms: 2

SUMMARY:
The purpose of this study is to determine wether autologous bone graft from iliac crest enhances bone union of tibial osteotomies, in the treatment of varus knee deformity.

DETAILED DESCRIPTION:
Opening-Wedge High Tibial Osteotomy is a classic procedure,but the use of autologous bone graft from iliac crest causes pain and bleeding. Bone union occur even without bone graft, but no clinical trials compared results of the twoo procedures.

ELIGIBILITY:
Inclusion Criteria:

* varus knee deformity
* unicompartmental arthrosis

Exclusion Criteria:

* patellar arthrosis
* lateral arthrosis
* inflammatory diseases
* bone healing impair drugs or diseases

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2006-04; Primary Completion 2008-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Clinical based bone union time | after 8 weeks

SECONDARY OUTCOMES:
X-ray femoro-tibial angle | 6 months, 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro R Zorzi, MD, Principal Investigator — University of Campinas, Brazil; João B Miranda, MD, PhD, Study Chair — University of Campinas, Brazil
Locations (1):
- Departamento de Ortopedia do Hospital de Clínicas da Unicamp, Campinas, São Paulo, Brazil